CLINICAL TRIAL: NCT01047709
Title: Positional Therapy After Stroke
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Devin Brown, Associate Professor, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: U024133
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Results first posted 2013-06-10 (Estimated); Last update posted 2013-06-10 (Estimated); Status verified 2013-06

CONDITIONS: Sleep Apnea; Stroke
MeSH Terms: conditions — Sleep Apnea Syndromes; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- positional therapy (Experimental): Avoidance of supine positioning.
  Interventions: Device: Positional therapy including the use of a special pillow
- Control (No Intervention): Position ad lib.

INTERVENTIONS:
Device: Positional therapy including the use of a special pillow — Avoidance of supine sleep via a special pillow and other measures.
  Other Names: Sona Pillow.
  Arms: positional therapy

SUMMARY:
Stroke is the leading cause of adult disability and the third leading cause of death in the United States. Unfortunately, there are few therapies that have been proven to improve stroke outcome. Sleep apnea is an emerging stroke risk factor and has a well established association with higher mortality and poor functional outcome following stroke. Over half of acute stroke patients have sleep apnea, suggesting that it may be a important target for therapy. Attenuation of sleep apnea severity may result in improved stroke outcomes. However, the standard treatment for sleep apnea is not well-tolerated among stroke patients. An alternative treatment is avoidance of supine sleep. Supine sleep is very common in acute stroke patients, and therefore this treatment may have particular relevance to the stroke population. The proposed study will be conducted in two phases. The first phase is a randomized, crossover design in which acute stroke patients will be given positional treatment (to avoid supine sleep) on one night during their stroke hospitalization. This will be compared with another night of sleeping without positional therapy. The order of treatments (standard vs positional therapy) will be random. The first phase will demonstrate the proof of concept: that stroke patients given positional therapy to avoid supine sleep will (1) sleep less on their backs, and (2) will have improved sleep apnea parameters with positional therapy. In the second phase, those identified to have sleep apnea will be randomized to receive positional therapy at home for three months, or standard therapy. This second phase will demonstrate the adherence/feasibility of three months of positional therapy, and will allow us to estimate effect size based on a functional outcome measure. The data obtained from this pilot clinical trial are essential to plan a large efficacy study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Probable ischemic stroke within prior 14 days

Exclusion Criteria:

* Any medical condition precluding the avoidance of supine posture or dictating the need for a particular position.
* Current use of CPAP (or other PAP), mechanical ventilation, or supplemental oxygen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-12; Primary Completion 2010-02 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Devin L Brown, MD, MS, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Svatikova A, Chervin RD, Wing JJ, Sanchez BN, Migda EM, Brown DL. Positional therapy in ischemic stroke patients with obstructive sleep apnea. Sleep Med. 2011 Mar;12(3):262-6. doi: 10.1016/j.sleep.2010.12.008. PMID 21306949

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a crossover study. One night with positional therapy (intervention) and one night of sleeping ad lib (control). The order was randomly assigned. Subjects were enrolled between 12/2008 and 2/2010.
Groups:
- Positional Therapy Night First, Then Control Night: Avoidance of supine positioning on the first night, followed by a second night of positioning ad lib.
- Control Night First, Then Positional Therapy Night: Position ad lib for the first night, then one night of avoidance of supine positioning.
Period: Positional Therapy (1 Night)
Arm/Group | Positional Therapy Night First, Then Control Night | Control Night First, Then Positional Therapy Night
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0
Period: Control/Positioning ad Lib (1 Night)
Arm/Group | Positional Therapy Night First, Then Control Night | Control Night First, Then Positional Therapy Night
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All study participants.
Arm/Group | All Study Participants
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 7
Age Continuous [Mean (Standard Deviation); unit: years] | 59 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Apnea-hypopnea Index
Description: Apnea-hypopnea index (AHI) is the sum of the apneas and hypopneas and divided by the hours of presumed sleep. AHI values are typically categorized as 5-15/hr = mild; 15-30/hr = moderate; and >= 30/h = severe. The relative treatment effect on AHI using GEE modeling.
Time Frame: 1 day
Measure: Median (Inter-Quartile Range); unit: events/hr
Groups:
- Positional Therapy Night: Avoidance of supine positioning.
- Control Night: Position ad lib
Arm/Group | Positional Therapy Night | Control Night
Number analyzed (Participants) | 18 | 18
events/hr | 27 [22 to 47] | 39 [21 to 54]
Statistical Analysis 1: Comparison: Positional Therapy Night vs Control Night; Relative treatment effect on AHI, using GEE modeling, accounting for crossover design; Test type: Superiority or Other; p = 0.011, GEE; relative % difference = 19.5, 95% CI 2-sided [4.9 to 31.9], Standard Deviation 23 — SD of control night
Statistical Analysis 2: Comparison: Positional Therapy Night vs Control Night; Relative treatment effect on AHI, using GEE modeling, accounting for crossover design; Test type: Superiority or Other; p = 0.011, GEE; Relative % difference = 19.5, 95% CI [4.9 to 31.9], Standard Deviation 16 — SD of intervention night

ADVERSE EVENTS:
Arm/Group | Positional Therapy Night | Control Night
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No